CLINICAL TRIAL: NCT00409201
Title: Phase 1 Study of Reboxetine Adjuvant Therapy and Cognitive and Behavioral Measures
Brief Title: Reboxetine Adjuvant Therapy for the Treatment of Schizophrenia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abarbanel Mental Health Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 284
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; reboxetine; cognitive; behavior
MeSH Terms: conditions — Schizophrenia; Behavior

INTERVENTIONS:
Drug: reboxetine adjuvant therapy

SUMMARY:
30 patients will randomly be selected and will be administered either reboxetine or a placebo. changes in cognition and behavior will be assessed by computer tests and scales during a six week study period.

DETAILED DESCRIPTION:
all participants will be administered panss, sans, esrs, calgary, progesterom, sexual functioning scale, ham-a, covy, hamilton depression scale, and cgi and cgi improved rating on the first visit, as well as blood tests, ecg and weight. they will then be tested using a computer cognitive test (cogscan test) that lasts about 45 minutes. next, they will be given either a two week dose of placebo or treatment (2 mg * 2 daily for first week, then 4 mg. day, 2 mg. night for the second week). after two weeks they the dose is increased to 4 mg. * 2 daily. at four weeks all tests are readministered, as well as at six weeks. the study is concluded at 6 weeks, following a readministration of tests. physical examination is also administered at the conclusion.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia all types
* 18>

Exclusion Criteria:

* uti
* >65
* non organic state
* no depression treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-03; Study Completion 2006-11

PRIMARY OUTCOMES:
sans, panss, hamilton, ham-a, calgary, physical examination, cogscan test

SECONDARY OUTCOMES:
esrs, progesterom, sexual functioning, covy, cgi, cgi improved

CONTACTS AND LOCATIONS:
Overall Officials: stanislav baranchik, md, Principal Investigator — abarbanel mhc
Locations (1):
- Abarbanel Medical Mental Health Center, Bat Yam, Israel

REFERENCES:
- [Background] Schutz G, Berk M. Reboxetine add on therapy to haloperidol in the treatment of schizophrenia: a preliminary double-blind randomized placebo-controlled study. Int Clin Psychopharmacol. 2001 Sep;16(5):275-8. doi: 10.1097/00004850-200109000-00004. PMID 11552770